CLINICAL TRIAL: NCT03544554
Title: The Effect of a Counseling and Training Program on the Treatment of Women With Overactive Bladder
Brief Title: Training and Counseling Program for Overactive Bladder Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Gulsen Cayir, Assistant professor, PhD, Biruni University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0925-0586
Record Dates: First submitted 2018-04-13; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder; healthy lifestyle behaviors; quality of life
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: The study sample included 100women (50 for the intervention and 50 for the control group) diagnosed with OAB syndrome. The control group was not provided with training. In addition to the pharmacological treatment, the intervention group was provided with a counseling and training program that consisted of a 45minute presentation based on Pender's Health Promotion Model. They were also given "A Manual for Training on HealthyLifestyleBehaviors among women with OAB". The intervention group was requested to follow a weekly-scheduled bladder training program, keep records on the Urinary Diary form for six weeks. In the first interview and in the third month, the women in the intervention and control groups were administered the Introductory Information Form, Urinary Diary (4day), 24hour Standard Pad Test, OAB-V8, King'sHealthQuestionnaire, Healthy LifestyleBehaviorScaleII, and BriefSymptomInventory. In addition, an Inspection Form was administered in the third month.
Masking Description: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group and control group (Experimental): This research is planned with semi experimental design
  Interventions: Behavioral: a counseling and training program that consisted of a 45-minute presentation based on Pender's Health Promotion Model. Within the scope of the counseling and training program

INTERVENTIONS:
Behavioral: a counseling and training program that consisted of a 45-minute presentation based on Pender's Health Promotion Model. Within the scope of the counseling and training program — The intervention group was provided with a counseling and training program that consisted of a 45-minute presentation based on Pender's Health Promotion Model.
  Other Names: The control group was not provided with training

SUMMARY:
The study concluded that HLSB training reduced OAB symptoms among women, improved the quality of their lives, changed their HLSBs, and positively affected their mental states. Thus, a holistic approach to the treatment of women with OAB increased the success of the treatment.

DETAILED DESCRIPTION:
The population of this study included all women who received treatment in the Urogynecology Outpatient Clinic of the Gynecology and Obstetrics Department in İstanbul Faculty of Medicine at İstanbul University between January 2015 and October 2016. Permission was obtained for the study from the Ethics Committee of İstanbul University Cerrahpaşa Faculty of Medicine and İstanbul University İstanbul Faculty of Medicine. The study sample included 100 women diagnosed with OAB syndrome. Of them, 50 were selected for the intervention group and 50 were selected for the control group.

Detailed information was given to the women beginning pharmacological treatment who met the inclusion criteria, and their consent was obtained using an Informed Voluntary Consent Form. During the pharmacological treatment, anticholinergic drugs, which contained active ingredients such as tolterodine 4 mg/day, trospium cl 60 mg/day, fesoterodine 4-8 mg/day, and solifenacin 5 or 10 mg/day were prescribed. The women in each group were instructed to take the prescribed anticholinergic drugs regularly, informed about the side effects of these drugs, and advised on the situations when they should seek immediate treatment before their next scheduled appointment. The women with OAB were divided into groups using random allocation (by drawing lots). To set an equal distribution of patients into the intervention and control groups, the group of the first patient was determined by lot, and the next patient was allocated to the other group.

The control group was not provided with training. In addition to the pharmacological treatment, the intervention group was provided with a counseling and training program that consisted of a 45-minute presentation based on Pender's Health Promotion Model. Within the scope of the counseling and training program, the patients were given information about the female reproductive system, anatomy and physiology of the urinary system, OAB definition, OAB symptoms, and HLSBs (adequate fluid intake, diet, prevention methods for urinary tract infections, weight control, regular bowel movements, smoking cessation, treatment of chronic diseases, and regular medication). The patients were informed about the importance of concentration, learning about pelvic floor muscle contraction and exercises and performing them regularly, as well as designing bladder training programs and sticking to them to manage urgency and urinary incontinence. They were also given "A Manual for Training on Healthy Lifestyle Behaviors among Women with Overactive Bladder". Figure 1 shows the HLSB development based on Pender's Health Promotion Model in OAB treatment.

The intervention group was requested to follow a weekly-scheduled bladder training program, keep records on the Urinary Diary form for six weeks, and bring this form at the end of each week. The researcher called each patient 8-10 times: every week during the first six weeks and once a month afterwards to encourage implementation of the practices for three months starting from the first interview. During the phone calls, the patients were asked about their drug use, average daily fluid intake, and any concerns as well as state of performing pelvic floor muscle contraction and exercises, sticking to the scheduled bladder training hours, and weight loss. The data obtained through these calls were recorded on the Practice Registration Form. The control group, on the other hand, was called once a month and instructed to continue taking their drugs, which was also recorded on the form.

In the first interview and in the third month, the women in the intervention and control groups were administered the Introductory Information Form, Urinary Diary (4-day), 24-hour Standard Pad Test, Overactive Bladder Questionnaire (OAB V8), King's Health Questionnaire (KHQ), Healthy Lifestyle Behavior Scale II (HLSB II), and Brief Symptom Inventory (BSI). In addition, an Inspection Form was administered in the third month.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Being literate
* Diagnosed with OAB
* Beginning to receive pharmacological treatment for OAB
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of a perceptual or psychiatric disorder which prevents communicating
* Presence of a neurological disorder
* Presence of neurological neuropathy caused by Diabetes Mellitus
* Second or higher stage pelvic organ prolapse
* Having an anti-incontinence surgery
* Being pregnant

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Overactive Bladder Questionnaire (OAB-V8) scores at 12 weeks | Intervention and control group cases were assessed at baseline and week 12. The OAB-v8 is a patient-reported outcome questionnaire which have six point rating system (0-40 scores).
  12 weeks a between implementation of pre-post test
Change from baseline King's Health Questionnaire (KHQ) scores at 12 weeks | Intervention and control group cases were assessed at baseline and week 12. KHQ is a patient self-administered self-report . The responses in KHQ have four point rating system. The eight subscales scored between 0 (best) and 100 (worst).
  12 weeks a between implementation of pre-post test.
Change from baseline Brief Symptom Inventory (BSI) scores at 12 weeks | Intervention and control group cases were assessed at baseline and week 12. The Brief Symptom Inventory (BSI) is a brief form of the Symptom Checklist, The responses in BSI have five point rating system(0-212 scores).
  12 weeks a between implementation of pre-post test
Change from baseline Healthy Life Style Behavior Scale II (HLSB II) scores at 12 weeks | Intervention and control group cases were assessed at baseline and week 12. HLSB II is used to measure the degree of engagement in a health-promoting lifestyle along 6 dimensions. The responses in HLPS II have four point rating system(52-208 scores).
  12 weeks a between implementation of pre-post test

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cayir G, Kizilkaya Beji N. The effect of a counseling and training program on the treatment of women with overactive bladder. Psychol Health Med. 2022 Sep;27(8):1726-1738. doi: 10.1080/13548506.2021.1916962. Epub 2021 Apr 19. PMID 33870822